CLINICAL TRIAL: NCT04983147
Title: The Effect of Training Given to Women With Obesity Patients According to the Health Belief Model on Obesity Beliefs and Obesity Management December,2018
Brief Title: The Effect of Training Given to Women With Obesity Patients According to the Health Belief Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Suheyla YARALI, Research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: sefa6192
Record Dates: First submitted 2021-05-12; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- health belief model based training manuel (Experimental): A training manual entitled "Do Not Stay Silent Towards Obesity" was prepared by the researcher to guide women in obesity management by affecting their beliefs on obesity in a positive way.
  Interventions: Other: Obesity Training Based on Health Belief Model
- powerpoint presentation with computer (Experimental): The presentation prepared based on the Health belief model was used in group training.
  Interventions: Other: Obesity Training Based on Health Belief Model
- video for obesity based on health beliefs (Experimental): In the literature; It is explained that the educator's use of representations such as video is more effective than verbal expression and reading, and facilitates learning both by hearing and seeing.For this reason, videos that will create awareness about the subject in the trainings were prepared by the researcher and used in the trainings.
  Interventions: Other: Obesity Training Based on Health Belief Model
- successful patients in obesity management (Experimental): Real-life stories of people who could manage obesity before and thought themselves healthier compared to their previous condition were shared with the group. People were invited to the trainings who had obesity before and managed to lose weight and trainings were given in the affective field.
  Interventions: Other: Obesity Training Based on Health Belief Model
- Post-training follow-up (Experimental): After the trainings given to women were completed, women were included in the follow-up program.For 6 mounts. This application will only be made in the experimental group.
  This follow-up will increase motivation and answer questions regarding obesity management.
  It was made by calling every 15 days.It will be made by phone call.
  Interventions: Other: Post-training follow-up

INTERVENTIONS:
Other: Obesity Training Based on Health Belief Model — Trainig was given with initiatives for cognitive and affective learning areas within the framework of health belief model.7 weeks.This application will only be made in the experimental group.
  Arms: health belief model based training manuel; powerpoint presentation with computer; successful patients in obesity management; video for obesity based on health beliefs
Other: Post-training follow-up — After 7 weeks of training to women were completed, women were included in the follow-up program.For 6 mounts. This application will only be made in the experimental group.It will be made by phone call.
  This follow-up will increase motivation and answer questions regarding obesity management.
  It was made by calling every 15 days.
  Arms: Post-training follow-up

SUMMARY:
This study was conducted to examine the effectiveness of the training provided to women with obesity based on the Health Belief Model on women's beliefs regarding obesity and obesity management of the women. Study population included 18 to 65 years old women with obesity and the study sample included 128 women (64 in the control group and 64 in the experimental group) determined by power analysis. Randomized controlled, single-blind clinical study included a total of 128 obesity woman

DETAILED DESCRIPTION:
Research data were collected by the researcher in the community health center. Research data were completed in 4 months. women in the experimental and control groups in collecting test data; Introductory Features consisting of 15 questions The form, which includes the Obesity health belief model scale and anthropometric measurements, was applied.Interventions were made on the women in the experimental situation, and no intervention was made on the control group.

Health Belief Model Scale in Obesity evaluates beliefs and attitudes towards. The scale consisting of 32 items in total The cronbach alpha coefficient is 0.80. Health Belief Model Scale in Obesity , sensitivity, seriousness, benefit and five sub-dimensions that can be used independently of each other, including perception of disability The importance of health; the level of importance individuals give to their health shows and consists of eight items (1, 2, 3, 4, 5, 6, 7, 8). Perceived sensitivity; health problems and complications that may develop due to obesity. to what level they find themselves susceptible, and the interventions to be made for obesity. evaluates at what level they find useful, and takes four items (12, 13, 14, 16) consists of. Perceived seriousness; To what extent do individuals have obesity and consists of four items (9, 10, 11, 17). Perceived benefit; what individuals gain in terms of their health when they manage obesity shows the level of awareness of the benefits and consists of 8 items (21, 22, 24, 25, 26, 27, 28, 32). Perceived obstacle; people's health recommendations for obesity. shows the level of the obstacles they perceive in practice and (15, 18, 19, 20, 23, 29, 30, 31).

The scale is a 5-point Likert type scale for each item. The importance of health in scale sub for the size; 1 for "Never", 2 for "Sometimes", 3 for "Frequently", 4 for "Very often", "Every evaluation is made by giving 5 points for "time". Perceived sensitivity, seriousness, obstacle and for perceptions of benefit; By giving 1 points for "absolutely disagree", 2 for "disagree", 3 for "indecisive", 4 for "agree", 5 for "absolutely agree" evaluation is done. total scale point average is not calculated. Each sub of the scale The scores of the items belonging to the subscale of the subscale are summed up and the number of items in each subscale is calculated. is divided. If every item in the scale was not answered, the number of items answered the corresponding ratings are summed up and the responses on that subscale are divided by the number of items. Sensitivity perception: Women see obesity as a disease and The definition of obesity in the educational content, how is it is evaluated and why it is an important health problem. Towards the perception of seriousness: Women should consider obesity as a serious health problem.

After evaluating the visual conditions, the educational content caused by obesity Health problems such as physical and mental illnesses are included. For the perception of benefit: It is important for women to manage obesity well. After evaluating the usefulness of the educational content, obesity health benefits of obesity management, proper nutrition and physical The benefits of the activity are included. Barrier perception: Perceived barriers by women in managing obesity After evaluating the obstacles encountered in managing obesity in the educational content what happened was discussed with the group, the things that could be done to overcome these obstacles were listed. education that includes the ability of women to manage obesity using appropriate ways For the perception of barriers: Perceived barriers by women in managing obesity After evaluating the obstacles encountered in managing obesity in the educational content what happened was discussed with the group, the things that could be done to overcome these obstacles were listed. education that includes the ability of women to manage obesity using appropriate ways program has been created. İmportance of health in scale, perceived usefulness, perceived the increase in the mean scores of the sensitivity and perceived seriousness sub-dimensions, The decrease in the average score of the perceived disability sub-dimension indicates that the applied training yields a positive result. Weight measurements of women, by placing the scales on a flat surface without slope, his thick clothes and shoes were removed, and it was made upright without moving.his thick clothes and shoes were removed, and it was built upright without moving.Women's height measurements with feet united and on the frankfort plane (head the angle between the neck and the neck is 90 degrees)Women's waist circumference measurements should be kept on a flat surface and excessive pressure by keeping the tape measure. hands and arms at both sides, feet close to each other (12-15 cm near) and the weight is evenly distributed on two feet from the belly button level. measured. A decrease in height, weight and BMI indicates that training is effective IMPACT STATEMENT What is already known on this subject? Behavior change is an important factor in obesity What the results of this study add? There are behavioral change initiatives by providing training, but by integrating the model use and training areas into the model, providing behavioral and attitude change will provide more effective and sustainable lifestyle changes in obesity.

What the implications are of these findings for clinical practice and/or further research? Studies about obesity patients, it is recommended that nursing interventions be carried out within the framework of models, and their training should be aimed at cognitive, affective and psychomotor areas and applied to different groups.In studies to be intended for obesity patients, it is recommended that nursing interventions be carried out within the framework of models, and their training should be aimed at cognitive, affective and psychomotor areas and applied to different groups. Its use in the Health belief model-based of obese with chronic diseases also contributes to disease. Health belief model-based training to be given to healthy individuals will contribute to the prevention of obesity.

ELIGIBILITY:
Inclusion Criteria:

* women with a waist circumference ≥88 cm
* with no previous training regarding obesity
* being at least a primary school graduate
* having no chronic diseases or mental or psychological disability limiting daily life activities

Exclusion Criteria:

* having an obesity surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form (questionnaire) | up to 12 weeks
  An introductory information form prepared by the researcher based on relevant literature was filled out by participants it included 15 questions regarding the age, marital status, family type, education status, social security, profession, income, and having children, doing exercise previously, the reason for quitting exercise, seeing a dietician and following a prescribed diet, and if so, the reason for abandoning the diet.
Health Belief Model Scale in Obesity (questionnaire-scale) | up to 12 weeks
  It is a questionnaire used as a measurement tool. Its validity and reliability have been proven. individuals to lose weight evaluate their beliefs and attitudes towards The scale consists of 32 items in total.
  The cronbach alpha coefficient is 0.80. health belief, sensitivity, seriousness, benefit and five sub-dimensions that can be used independently of each other, including the perception of obstacles exists.The scale is a 5-point Likert type scale for each item. The total scale score average of the survey is not calculated. Each sub-scale The scores of the items belonging to the sub-scale of the scale are calculated by adding up. If each item in the scale is not answered, the number of items answered The corresponding ratings are calculated by summing, and the responses on that subscale are calculated.
  divided by the number of items.
Health Belief Model Scale in Obesity-Importance of Health (questionnaire-scale) | up to 12 weeks
  The importance of health; the level of importance individuals give to their health and consists of eight items (1, 2, 3, 4, 5, 6, 7, 8). The higher the score, the higher the health level.
Health Belief Model Scale in Obesity- Perceived sensitivity (questionnaire-scale) | up to 12 weeks
  Perceived sensitivity; health problems and complications that may develop due to obesity. at what level they find themselves susceptible, and interventions for obesity evaluate what level they find useful and choose from four items (12, 13, 14, 16).
  consists of. The higher the score, the higher the sensitivity level.
Health Belief Model Scale in Obesity- Perceived severity (questionnaire-scale) | up to 12 weeks
  Perceived seriousness; At what level do individuals consider obesity a serious disease? evaluates what they see as their own and consists of four items (9, 10, 11, 17).
Health Belief Model Scale in Obesity- Perceived benefit (questionnaire-scale) | up to 12 weeks
  Perceived benefit; what individuals gain in terms of their health when they manage obesity shows the level of awareness of the benefits and consists of 8 items (21, 22, 24, 25, 26, 27, 28, 32). As the score increases, the level of perception increases as a benefit.
Health Belief Model Scale in Obesity- Perceived barrier (questionnaire-scale) | up to 12 weeks
  Perceived barrier; health recommendations of individuals for obesity. It shows the level of barriers they perceive in practice and consists of eight items.
  (15, 18, 19, 20, 23, 29, 30, 31).It is understood that as the perceived obstacle score decreases, the level of disability decreases.
Height Meter | up to 12 weeks
  Length Meter: SECA brand 20 - 207 cm capacity, height measurement with 1mm accuracy It is the length measuring stick that provides the opportunity.
weighing machine | up to 12 weeks
  weighing machine: SECA brand 200 kg capacity, 100 g precision weighing, wide and non-slip platform, large LCD number display scale.
body mass index calculation | up to 12 weeks
  weight and height will be combined to report BMI in kg/m^2 Weight assessment was made after the application. The change in body mass index was evaluated. It was determined whether women lost weight or not.

SECONDARY OUTCOMES:
Health Belief Model Scale in Obesity ((questionnaire-scale) | through study completion, an average of 1 year
  It is a questionnaire used as a measurement tool. Its validity and reliability have been proven. individuals to lose weight evaluate their beliefs and attitudes towards The scale consists of 32 items in total.
  The cronbach alpha coefficient is 0.80. health belief, sensitivity, seriousness, benefit and five sub-dimensions that can be used independently of each other, including the perception of obstacles exists.The scale is a 5-point Likert type scale for each item. The total scale score average of the survey is not calculated. Each sub-scale The scores of the items belonging to the sub-scale of the scale are calculated by adding up. If each item in the scale is not answered, the number of items answered The corresponding ratings are calculated by summing, and the responses on that subscale are calculated.
  divided by the number of items.
Health Belief Model Scale in Obesity-Importance of Health (questionnaire-scale) | through study completion, an average of 1 year
  The importance of health; the level of importance individuals give to their health and consists of eight items (1, 2, 3, 4, 5, 6, 7, 8). The higher the score, the higher the health level.
Health Belief Model Scale in Obesity- Perceived sensitivity (questionnaire-scale) | through study completion, an average of 1 year
  Perceived sensitivity; health problems and complications that may develop due to obesity. at what level they find themselves susceptible, and interventions for obesity evaluate what level they find useful and choose from four items (12, 13, 14, 16).
  consists of. The higher the score, the higher the sensitivity level.
Health Belief Model Scale in Obesity- Perceived severity (questionnaire-scale) | through study completion, an average of 1 year
  Perceived seriousness; At what level do individuals consider obesity a serious disease? evaluates what they see as their own and consists of four items (9, 10, 11, 17).
Health Belief Model Scale in Obesity- Perceived benefit (questionnaire-scale) | through study completion, an average of 1 year
  Perceived benefit; what individuals gain in terms of their health when they manage obesity shows the level of awareness of the benefits and consists of 8 items (21, 22, 24, 25, 26, 27, 28, 32). As the score increases, the level of perception increases as a benefit.
Health Belief Model Scale in Obesity- Perceived barrier (questionnaire-scale) | through study completion, an average of 1 year
  Perceived barrier; health recommendations of individuals for obesity. It shows the level of barriers they perceive in practice and consists of eight items.
  (15, 18, 19, 20, 23, 29, 30, 31).It is understood that as the perceived obstacle score decreases, the level of disability decreases.
Height Meter | through study completion, an average of 1 year
  Length Meter: It measures the height of the individual. SECA brand 20 - 207 cm capacity, height measurement with 1mm accuracy It is the length measuring stick that provides the opportunity.
weighing machine | through study completion, an average of 1 year
  weighing machine: SECA brand 200 kg capacity, 100 g precision weighing, wide and non-slip platform, large LCD number display scale.
body mass index calculation | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2 Weight assessment was made after the application. The change in body mass index was evaluated. It was determined whether women lost weight or not.

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Yaralı, Principal Investigator — Study Principal Investigator
Locations (1):
- Süheyla Yaralı, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No